CLINICAL TRIAL: NCT05616416
Title: Institute of Sciences in Emergency Medicine - International Big Data Centre in Emergency Medicine
Brief Title: International Big Data Centre in Emergency Medicine
Status: Recruiting | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Abdelouahab Bellou, Director of Institute of Sciences in Emergency Medicine, Guangdong Provincial People's Hospital
Other Study IDs: KY-N-2022-105-01
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Emergency Medicine
Keywords: Machine Learning; Data Mining; Artificial Intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All ED Patient: All patients visited the emergency department during the period.

SUMMARY:
This observational study aims to use electronic health records to build an International Big Data Centre in Emergency Medicine, within the Institute of Sciences in Emergency Medicine (ISEM) at the Guangdong Provincial People's Hospital. The main questions it seeks to answer are not limited to the following:

* Identify the relationship between Emergency Department Length of Stay (EDLOS), Mortality, and Adverse Events (AE)
* Identify the risk factors associated with high mortality and AE rate among patients who experience prolonged EDLOS
* Other research questions related to emergency medicine, such as building prediction and cluster models for acute diseases

DETAILED DESCRIPTION:
The relationship between the emergency department length-of-stay (EDLOS), mortality, and adverse events (AE) rate remains unclear and underestimated. EDLOS is the time elapsed between the time of arrival and the time of the release of a patient admitted to ED. Mortality is defined as short-term (14 hours, 48 hours, 7 days, 15 days) and 30 days death of patients managed in the ED discharged or admitted. An AE is an event that can result whether from medical mismanagement or happen by accident and causes physical and mental harm to the patient during the stay and remains after leaving. To separate the mismanagement from accidental causes i.e., compliant management but the unfortunate situation or persons, this study will refer to indicators that are objectively measurable and can be compared at different times throughout the patient's stay in the ED.

The hypothesis is that a prolonged stay of the patients in the ED especially without diagnosis or decision of admission is associated with increased mortality and AEs. This project will test this hypothesis through a prospective international multicenter study in contributing to whether a prolonged EDLOS is associated with an increased rate of adverse outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Every patient who ever visited Emergency Department from 2011-2022

Exclusion Criteria:

* Patients with missing demographic (age, gender, etc.) and triage data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be everybody who visited the Emergency Department.
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
In-hospital Mortality | From date of ED triage until the date of discharge or date of death from any cause, whichever came first, assessed up to 1 month
  IHM

SECONDARY OUTCOMES:
Number of Adverse Events | From date of ED triage until the date of discharge or date of death from any cause, whichever came first, assessed up to 1 month
  AE

CONTACTS AND LOCATIONS:
Overall Officials: Abdelouahab Bellou, MD, PhD, MSc, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided